CLINICAL TRIAL: NCT05194358
Title: Phase 1, Open Label, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Stabilized Isoamyl Nitrite (SIAN) Nasal Spray in Healthy Adults
Brief Title: Study of SIAN Nasal Spray in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EBS-SIN-001
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cyanide Poisoning
Keywords: Cyanide Exposure; Cyanide; Stabilized Isoamyl Nitrite (SIAN); Isoamyl Nitrite (IAN)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 SIAN (Experimental): SIAN dose of 0.28 mg/kg (20 μL) will be administered from a single syringe-based spray device into left nostril.
  Interventions: Drug: Stabilized Isoamyl Nitrite (SIAN)
- Cohort 2 SIAN (Experimental): SIAN dose of 0.73 mg/kg (50 μL) will be administered from a single syringe-based spray device into left nostril.
  Interventions: Drug: Stabilized Isoamyl Nitrite (SIAN)
- Cohort 3 SIAN (Experimental): SIAN dose of 1.45 mg/kg (100 μL) will be administered from a single syringe-based spray device into left nostril.
  Interventions: Drug: Stabilized Isoamyl Nitrite (SIAN)
- Cohort 4 SIAN (Experimental): SIAN dose of 2.18 mg/kg (150 μL) will be administered from a single syringe-based spray device into left nostril.
  Interventions: Drug: Stabilized Isoamyl Nitrite (SIAN)
- Cohort 5 SIAN (Experimental): SIAN dose of 2.90 mg/kg (200 μL) will be administered in two syringe-based spray devices, each containing 100 μL, with dose administered in left then right nostril, one device per nostril.
  For doses of 2.90 milligram/kilogram (200 microliter) and higher, the dose will be split equally between the two nostrils to avoid drug overflow from the nose (using two syringe-based spray devices one immediately followed by the other). Lower doses will be administered by a single device to one nostril.
  Interventions: Drug: Stabilized Isoamyl Nitrite (SIAN)
- Cohort 6 SIAN (Experimental): SIAN dose of 3.63 mg/kg (250 μL) will be administered in two syringe-based spray devices, each containing 125 μL, with dose administered in left then right nostril, one device per nostril.
  Interventions: Drug: Stabilized Isoamyl Nitrite (SIAN)
- Cohort 7 SIAN (Experimental): SIAN dose of 4.35 mg/kg (300 μL) will be administered in two syringe-based spray devices, each containing 150 μL, with dose administered in left then right nostril, one device per nostril.
  Interventions: Drug: Stabilized Isoamyl Nitrite (SIAN)

INTERVENTIONS:
Drug: Stabilized Isoamyl Nitrite (SIAN) — SIAN is comprised of isoamyl nitrite (IAN) stabilized with 4% by weight epoxidized linseed oil (ELSO) and administered by intranasal (IN) delivery as a nasal spray.
  A syringe-based spray device will be used to administer the SIAN product. This syringe-based spray device, consists of a Hamilton type syringe connected to a tip that functions as an atomizer, to provide an optimal spray plume for nasal absorption while minimizing exposure to lungs.

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single ascending doses of Stabilized Isoamyl Nitrite (SIAN) nasal spray in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1, open label, single ascending dose (SAD) study of Stabilized Isoamyl Nitrite (SIAN) nasal spray to assess safety, PK and PD.

The study will consist of seven cohorts, with up to 10 subjects planned per cohort, for a total of 70 subjects. Each cohort will include 10 healthy male or non-pregnant female subjects, aged 18 to 45 years inclusive. There will be a screening period from Day -28 to Day -2 for all study subjects. Subjects will stay overnight at the site the day prior to dosing (Day -1) and the day of dosing (Day 1). They will be evaluated until 24 hours after dosing (Day 2) prior to discharge from the phase 1 clinic. Subjects will return for an End of Study Visit at Day 8 after dosing.

Within cohorts one and two, the first two subjects will be dosed as sentinels, while cohorts three to seven will dose the first three subjects as sentinels. Upon completion of the Day 8 (end of study/early withdrawal) visit, safety data, including clinical and laboratory data, and raw PD/PK data will be reviewed by the Principal Investigator (PI) and Medical Monitor (MM) and Safety Monitoring Committee (SMC). If exposure is evident based on raw IAA PK data and PD response signals are detected, the remaining subjects (eight subjects for cohorts one and two and seven subjects for cohorts three to seven) will be dosed. If no exposure and/or PD response signals are detected during sentinel dosing, escalation to the next cohort may be permitted by the SMC.

For cohorts where all 10 subjects are dosed, the SMC will review the entire cohort data through each subject's Day 8 visit and provide a recommendation on either, (a) dose escalation to the next cohort, (b) lowering the next dose level, or (c) stopping enrollment based on dose-limiting toxicity.

Each new cohort will be dosed following the same procedure as the prior cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent (and assent as applicable) voluntarily signed by subject/guardian/legally acceptable representative.
2. Generally healthy, in the opinion of the PI, medical history, physical examination, vital signs, ECG and laboratory assessments at Screening.
3. Male or non-pregnant female.
4. Aged 18-45 years, inclusive, at the time of informed consent.
5. Have adequate venous access for phlebotomies.
6. For Women who are EITHER A or B:

   A. Not of childbearing potential: surgically sterile (at least six weeks post bilateral tubal ligation, bilateral oophorectomy or hysterectomy); or post-menopausal (defined as ≥50 years of age with a history of ≥12 consecutive months without menses prior to randomization in the absence of other pathologic or physiologic causes and screening follicle-stimulating hormone [FSH] > 30 mIU/mL)

   B. Women of childbearing potential who are not planning to be pregnant during the study period and who meet criteria i - iv: i. Negative serum pregnancy test at Screening Visit ii. Negative urine pregnancy test prior to dosing at Day -1 (Baseline) iii. Not currently breastfeeding iv. Using one of the following highly effective methods of contraception during the study period:
   * Combined estrogen and progestogen, or progestogen-only hormonal contraception associated with inhibition of ovulation (e.g. implants, pills, patches) initiated ≥30 days prior to Day 1
   * Intrauterine device (IUD) inserted ≥30 days prior to Day 1
   * Double barrier type of birth control (e.g. female condom, diaphragm or cervical cap and spermicidal foam/gel/cream/suppository, or male condom with diaphragm, male condom with cervical cap)
7. Body mass index (BMI) between 18 and 34 kg/m2, inclusive.

Exclusion Criteria:

1. Acute disease not resolved at least 4 weeks before Baseline (Day -1).
2. Any chronic clinical condition that requires active treatment of any kind. However, subjects that are on thyroid hormone replacement therapy are eligible if clinically euthyroid and on a stable dose of thyroxine for at least 2 years.
3. Medical history of cardiovascular (including symptomatic or asymptomatic aortic or mitral valvular disease, hypertension), renal, pulmonary and neurological conditions.
4. Active treatment for erectile dysfunction, continuous or on demand, within 4 weeks of baseline.
5. Orthostatic hypotension (at any time prior to dosing) or history of syncope of any cause.
6. Clinically significant ocular condition, other than a requirement for corrective lenses.
7. Any cancer other than the following:

   1. Any non-metastatic cancer (excluding hematologic malignancies) or melanoma of which the subject has been disease-free for at least five years; or
   2. Localized skin cancer that has been resected at least 4 weeks prior to Screening (including squamous cell and basal cell carcinomas).
8. History of intolerance to nitrites, nitrates or IAN and/or any of the study drug components (including ELSO (Epoxidized linseed oil)).
9. Contraindication to methylene blue as per the medical history of the subject.
10. History of nasal disorders, chronic sinusitis, sinonasal surgery including rhinoplasty, or significant abnormalities of the nasal anatomy including septum deviations.
11. Piercing of the nose that could interfere with study drug administration or absorption or study assessments, as judged by the investigator.
12. Participation in another clinical study and/or use of any drug, vaccine, device or combination product in the context of a clinical research study within 30 days prior to Baseline (Day -1) or administration of a biological product in the context of a clinical research study within 90 days prior to Baseline (Day -1).
13. Red blood cell G6PD (glucose-6-phosphate dehydrogenase) deficiency, by laboratory testing at Screening.
14. Any lab values outside the normal range that are deemed to be clinically significant in the PI and/or Medical Monitor's judgement.
15. Hemoglobin (Hb) < 12.0 g/dL for females or < 13.5 g/dL for males at Screening.
16. Methemoglobin > 3% at Screening or Day -1.
17. Any history or family history of congenital methemoglobinemia.
18. Has a positive serology test for human immunodeficiency virus antibodies, hepatitis B virus surface antigen or hepatitis C virus antibodies at Screening.
19. Any ECG assessment that is outside the normal range that is deemed clinically significant per the Principal Investigator's and/or Medical Monitor's judgement at Screening or Day -1 ECG; however, abnormal readings for the following benign conditions will be acceptable for inclusion in the study: early repolarization, nonspecific ST-T wave pattern or changes, right axis deviation (axis ≤ 110°), first degree atrioventricular block (PR interval < 240 millisecond (ms)), nonspecific intraventricular conduction delay (QRS < 120 ms), indeterminate axis and short PR interval (no delta wave present). On standard 12-lead ECG, a QTcF interval of >450 ms for males and >470 for females. If a single ECG QTcF is >450 ms for males and >470 for females, two more ECGs will be obtained over a 5-10 min period and the average of the QTcF interval from the 3 ECGs readings will be used to determine eligibility.
20. Any scheduled or anticipated medical intervention or surgical procedure, including dental procedures, during study participation, from Screening through Day 8.
21. History of chronic or current tobacco use. Subjects with more than 10 years of tobacco cessation might be included if they are considered healthy according to Investigator's opinion and medical history.
22. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]) or positive alcohol breath test at Screening or Day -1.
23. Positive test result on urine drug screen (cocaine, marijuana, phencyclidine, amphetamine, methamphetamine, opioids including methadone, ecstasy), any evidence of ongoing drug abuse or dependence (including alcohol), or recent history (over the past five years) of treatment for alcohol or drug abuse within 1 year prior to screening or positive standard urine drug test at Screening or Day -1.
24. History of the use of poppers, (alkyl nitrites) or positive standard urine drug screen.
25. Has donated plasma or blood or intends to donate within 30 days prior to Day 1 or during the course of the study.
26. Has received any medication, either prescription or non-prescription, including dietary supplements or herbal medications (e.g., quercetin, Gingko Biloba, palmetto, etc.), within 14 days or less than 5 half-lives prior to Baseline (Day -1) and is unable to refrain from any medication during study participation. If more than 5-half-lives is passed from the last dose of the over-the-counter medications listed in the protocol prior to admission Day-1, subjects will be eligible. The only allowed exception is hormonal birth control.
27. Psychological and/or emotional problems, which would render the informed consent invalid or limit the ability of the subject to comply with the study requirements.
28. Member or immediate family member of an investigative site or Sponsor team member.
29. Known lack of treatment compliance from prior studies or ongoing medical care based on medical records and Investigator's assessment.
30. Judged by the Investigator or Sponsor to be inappropriate/ineligible for the study for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Related Serious Adverse Events (SAEs) | Through Day 8
  Incidence of related SAEs
Methemoglobin (MetHb) level | Through 360 minutes post-dose
  To determine the dose that will result in a 6-10% MetHb level

SECONDARY OUTCOMES:
PK Endpoint: Maximum observed concentration (Cmax) of Isoamyl Alcohol (IAA metabolite) | Through 59 minutes post-dose
  Assess the maximum observed concentration (Cmax) of IAA
PK Endpoint: Time at which Cmax occurs (Tmax) of IAA | Through 59 minutes post-dose
  Assess the time at which Cmax occurs (Tmax) of IAA
PK Endpoint: Apparent first order terminal elimination half-life (t 1/2) of IAA | Through 59 minutes post-dose
  Assess the apparent first order terminal elimination half-life (t 1/2) of IAA
PK Endpoint: Area under the concentration-time curve from time 0 to 10 minutes post-dose (AUC 0-10min) of IAA | Through 59 minutes post-dose
  Assess the area under the concentration-time curve from time 0 to 10 minutes post-dose (AUC 0-10min) of IAA
PK Endpoint: Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC 0-last) of IAA | Through 59 minutes post-dose
  Assess the area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC 0-last) of IAA
PK Endpoint: AUC 0-t plus the additional area extrapolated to infinity (AUC 0-inf) of IAA | Through 59 minutes post-dose
  Assess the AUC 0-t plus the additional area extrapolated to infinity (AUC 0-inf) of IAA
PD Endpoint: Cmax of MetHb | Through 360 minutes post-dose
  Assess the Cmax of MetHb
PD Endpoint: AUC0-t of MetHb | Through 360 minutes post-dose
  Assess the AUC0-t of MetHb
PD Endpoint: t1/2 of MetHb | Through 360 minutes post-dose
  Assess the t1/2 of MetHb
PD Endpoint: The maximum change from baseline (Emax) of MetHb | Through 360 minutes post-dose
  Assess the maximum change from baseline (Emax) of MetHb
PD Endpoint: Time of reaching Emax (TEmax) of MetHb | Through 360 minutes post-dose
  Assess Time of reaching Emax (TEmax) of MetHb
PD Endpoint: Time to recovery to baseline values of MetHb | Through 360 minutes post-dose
  Assess the time to recovery to baseline values of MetHb
PD Endpoint: Area under the effect curve (AUEC(0-t)) of the fraction of MetHb (%) | Through 360 minutes post-dose
  Assess the area under the effect curve (AUEC(0-t)) of the fraction of MetHb (%)
PD Endpoint: for BP maximum change from baseline (Emax) | Through 8 hours post dose
  Assess the Emax for BP
PD Endpoint: for BP maximum change from TEmax | Through 8 hours post dose
  Assess the TEmax for BP
PD Endpoint: Time to recovery to baseline values for BP (mm Hg) | Through 8 hours post dose
  Assess the time to recovery to baseline values for BP (mm Hg)
PD Endpoint: Emax for SpO2 by pulse oximetry | Through 8 hours post dose
  Assess the Emax for SpO2
PD Endpoint: TEmax for SpO2 by pulse oximetry | Through 8 hours post dose
  Assess the TEmax for SpO2
PD Endpoint: Time to recovery to baseline SpO2 (%) | Through 8 hours post dose
  Assess the time to recovery to baseline SpO2 (%)
PD Endpoint: Emax for HR (heart rate) (beats/min) | Through 8 hours post dose
  Assess the Emax for HR (beats/min)
PD Endpoint: TEmax for HR (beats/min) | Through 8 hours post dose
  Assess the TEmax for HR (beats/min)
PD Endpoint: Time to recovery to baseline for HR (beats/min) | Through 8 hours post dose
  Assess the time to recovery to baseline for HR (beats/min)
Safety Endpoint: Adverse Events (AEs) | Through Day 8
  Incidence of AEs
Safety Endpoint: Toxicity grade 1 or higher of vital signs | Through Day 8
  Incidence of toxicity grade 1 or higher of vital signs
Safety Endpoint: Toxicity grade 1 or higher of clinical laboratories | Through Day 8
  Incidence of toxicity grade 1 or higher of clinical laboratories
Safety Endpoint: Orthostatic Hypotension | Through 60 minutes Post-Dose
  Incidence of orthostatic hypotension (drop in systolic blood pressure of at least 20 millimeters of mercury (mm Hg) or diastolic blood pressure of at least 10 mm Hg within three minutes of standing).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Austin Clinical Research Unit - PPD Phase I Clinic, Austin, Texas